CLINICAL TRIAL: NCT01617421
Title: Pilot Study of Yoga as Self-Care for Arthritis in Minority Communities
Brief Title: Yoga as Self-Care for Arthritis in Minority Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 120145; 12-CC-0145
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Results first posted 2019-07-01 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2018-04-17

CONDITIONS: Rheumatoid Arthritis; Arthritis
Keywords: Yoga; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Yoga

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Yoga (Experimental): This study used Hatha yoga (influenced by Integral, Iyengar, and Kripalu yoga) which includes postures (asanas), breathing techniques (pranayama) and meditation [9]. Biweekly, 60-minute, bilingual yoga classes were offered for 8 weeks at a yoga studio in Washington, DC. Classes were kept small (3-10 participants) to allow for pose modifications as needed for each participant. Participants were given instructions, bilingual manuals, and yoga equipment to encourage home practice. Participants were asked to keep journals to document the frequency and duration of home practice and their experience while on the study. After the last class, a yoga DVD and a list of local yoga studios were given to encourage continued practice.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: Yoga — This study used Hatha yoga (influenced by Integral, Iyengar, and Kripalu yoga) which includes postures (asanas), breathing techniques (pranayama) and meditation [9]. Biweekly, 60-minute, bilingual yoga classes were offered for 8 weeks at a yoga studio in Washington, DC. Classes were kept small (3-10 participants) to allow for pose modifications as needed for each participant. Participants were given instructions, bilingual manuals, and yoga equipment to encourage home practice. Participants were asked to keep journals to document the frequency and duration of home practice and their experience while on the study. After the last class, a yoga DVD and a list of local yoga studios were given to encourage continued practice.

SUMMARY:
Background:

* People with arthritis should be active. Regular exercise leads to less pain, more energy, improved sleep, and better day-to-day function. Yet arthritis is one of the most common reasons people give for limiting activities.
* Yoga for arthritis has been studied before. However, few studies have included minorities. Making changes to yoga classes based on language and culture may help people use yoga to care for their arthritis symptoms. Researchers want to see if minority populations with arthritis will come to and benefit from yoga classes.

Objectives:

- To see if yoga classes designed for people with arthritis will be acceptable to minorities with arthritis.

Eligibility:

* Adults at least 18 years of age who are enrolled in the Natural History of Rheumatic Disease in Minority Communities study.
* Participants will have osteoarthritis or rheumatoid arthritis.
* Participants will be able to speak and read English or Spanish.

Design:

* The total study period covers 10 weeks.
* The first study visit will include an initial questionnaire about health and arthritis. Participants will also have a physical exam.
* Participants will have yoga classes twice a week for 8 weeks. The classes will be 1 hour long each.
* After completing the yoga classes, participants will complete another questionnaire about their health. They will have a final physical exam.
* Follow-up contact will be made 3 months after the end of the study.

DETAILED DESCRIPTION:
Background:

Arthritis is the most common cause of disability, and is associated with activity limitation, work disability and significant health care costs. Approximately 50 million US adults have doctor-diagnosed arthritis. Non-Hispanic blacks and Hispanics have worse arthritis impact despite having the same or lower prevalence of arthritis compared to non-Hispanic whites. People with arthritis who exercise regularly have less pain, more energy, improved sleep and better day-to-day function. Yet, arthritis is one of the most common reasons for limiting physical activity. Improving health quality for people with chronic disease requires patients to take responsibility for their own care. Self-efficacy enhancing interventions may enable individuals to undertake self-care activities that improve physical and mental well-being. Attention is now being focused on complementary and integrated non-pharmacologic self-care approaches. Yoga is among the top 10 complementary and alternative medicine (CAM) modalities. Stretching, strength, posture, balance, and the ability to adjust pace and intensity are important safety components for patients with arthritis, all of which yoga encompasses. Mind-body interventions, such as yoga, that teach stress management with physical activity may be well suited for investigation in both osteoarthritis (OA) and rheumatoid arthritis (RA). Yoga users are predominately white, female, and college educated. In a descriptive study of patients enrolled in the Natural History of Rheumatic Disease in Minority Communities protocol only 4.6% were doing yoga. These disparities may be related to cost, access, and cultural beliefs. There are few studies that examine yoga in minority populations; none of these address arthritis.

Study Objective:

The primary objective of this study is to determine the feasibility and acceptability of providing yoga to an urban, minority population with arthritis.

Secondary Objective:

To determine the appropriateness of specific physical and psychosocial measures for this population, and intervention with a focus on physical function and patient reported measures.

Tertiary Objective:

To determine the feasibility of using computerized self-interview (with assistance) to capture baseline and final status.

Eligibility:

Adult patients (18 years or older) enrolled in the Natural History of Rheumatoid Disease in Minority Communities protocol with a diagnosis of osteoarthritis, rheumatoid arthritis or systemic lupus erythematosus (SLE).

Design:

A pilot study to evaluate the feasibility and acceptability of conducting a study based on a yoga intervention for arthritis in minority communities. Assessments will be made from a convenience sample of 20 RA/OA participants and 5 SLE participants undergoing an 8-week program of yoga classes consisting of 60-minute sessions, twice a week. The yoga classes are designed especially for people with arthritis.

ELIGIBILITY:
-

INCLUSION CRITERIA:

- Adult patients enrolled in the NIAMS Natural History of

Rheumatic Disease in Minority Communities

* Diagnosis of osteoarthritis (OA) or rheumatoid arthritis (RA)
* Willingness and ability to provide informed consent
* Age greater than or equal to 18 years

EXCLUSION CRITERIA:

* Recent (less than 6 months) or planned joint surgery
* Use of assistive ambulatory devices
* Other significant medical or psychiatric conditions, including other inflammatory conditions
* Hyper-mobility or unstable disease that could compromise participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-05-31; Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly R Middleton, R.N., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Middleton KR, Ward MM, Haaz S, Velummylum S, Fike A, Acevedo AT, Tataw-Ayuketah G, Dietz L, Mittleman BB, Wallen GR. A pilot study of yoga as self-care for arthritis in minority communities. Health Qual Life Outcomes. 2013 Apr 2;11:55. doi: 10.1186/1477-7525-11-55. PMID 23548052
- [Background] Middleton KR, Andrade R, Moonaz SH, Muhammad C, Wallen GR. Yoga Research and Spirituality: A Case Study Discussion. Int J Yoga Therap. 2015;25(1):33-5. doi: 10.17761/1531-2054-25.1.33. PMID 26667286
- [Background] Middleton KR, Haaz Moonaz S, Hasni SA, Magana Lopez M, Tataw-Ayuketah G, Farmer N, Wallen GR. Yoga for systemic lupus erythematosus (SLE): Clinician experiences and qualitative perspectives from students and yoga instructors living with SLE. Complement Ther Med. 2018 Dec;41:111-117. doi: 10.1016/j.ctim.2018.09.001. Epub 2018 Sep 8. PMID 30477826
- [Background] Middleton KR, Magana Lopez M, Haaz Moonaz S, Tataw-Ayuketah G, Ward MM, Wallen GR. A qualitative approach exploring the acceptability of yoga for minorities living with arthritis: 'Where are the people who look like me?'. Complement Ther Med. 2017 Apr;31:82-89. doi: 10.1016/j.ctim.2017.02.006. Epub 2017 Mar 1. PMID 28434476
- [Result] Middleton KR, Ward MM, Haaz Moonaz S, Magana Lopez M, Tataw-Ayuketah G, Yang L, Acevedo AT, Brandon Z, Wallen GR. Feasibility and assessment of outcome measures for yoga as self-care for minorities with arthritis: a pilot study. Pilot Feasibility Stud. 2018 Feb 20;4:53. doi: 10.1186/s40814-018-0248-x. eCollection 2018. PMID 29484197
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-CC-0145.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Yoga
Started | 18
Completed | 12
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Yoga
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 7
  More than one race | 1
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Self-Efficacy Exercise
Description: The Chronic Disease Self-Efficacy-Exercise Regularly Scale is a 3-item scale used to measure confidence in exercising regularly based on a Likert scale from 1 (not at all confident) to 10 (totally confident). The mean value was calculated based on participant responses to all three items.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga
Number analyzed (Participants) | 12
units on a scale | 6.1 [4.0 to 8.1]

2. Primary Outcome: Self-Efficacy Exercise
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga
Number analyzed (Participants) | 12
units on a scale | 7.5 [6.8 to 8.1]

3. Primary Outcome: Health-Promoting Lifestyle Profile II Score
Description: Health Promoting Lifestyle Profile (HPLP II) was used to measure the extent to which adults engage in a health-promoting lifestyle - Likert-type scales ranged from (1-never to 4-routinely). Subscales included: spiritual growth, interpersonal relations, nutrition, physical activity, health responsibility, and stress management. The mean value was calculated based on participant responses to all six subscales.
Time Frame: Baseline
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga
Number analyzed (Participants) | 12
units on a scale | 2.3 [2.0 to 2.6]

4. Primary Outcome: Health-Promoting Lifestyle Profile II Score
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Yoga
Number analyzed (Participants) | 12
units on a scale | 2.8 [2.5 to 3.1]

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Yoga
All-Cause Mortality (participants affected / at risk) | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Yoga (N=18)
Pain (General disorders) | 2 (2)
Discomfort (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As some patients experienced arthritis pain prior to participating in yoga study, it's not easy to differentiate between pre-existing arthritis pain symptoms and effects of yoga practice.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes